CLINICAL TRIAL: NCT04003389
Title: A Randomized, Placebo-Controlled, Double-Blind Phase 3 Clinical Study to Investigate the Long-Term Safety of Fezolinetant in Women Suffering From Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Find Out How Safe Long-term Treatment With Fezolinetant is in Women With Hot Flashes Going Through Menopause
Acronym: Skylight 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0304; 2019-000275-16 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Hot Flashes
Keywords: menopause; fezolinetant; ESN364; vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fezolinetant 30 mg (Experimental): Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, once daily (QD) for a period of 52 Weeks.
  Interventions: Drug: fezolinetant
- Fezolinetant 45 mg (Experimental): Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD for a period of 52 Weeks.
  Interventions: Drug: fezolinetant
- Placebo (Placebo Comparator): Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, QD for a of period of 52 Weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fezolinetant — administered orally
  Arms: Fezolinetant 30 mg; Fezolinetant 45 mg
Drug: placebo — administered orally
  Arms: Placebo

SUMMARY:
This study was for women in menopause with hot flashes. Menopause, a normal part of aging, was the time of a woman's last period. Hot flashes can interrupt a woman's daily life.

The purpose of this study was to find out how safe it is for these women to take fezolinetant in long term (up to 52 weeks). To do that, the study looked at the number and severity of the "adverse events." Those were the side effects that study participants had while they were in the study.

The study treatments were fezolinetant 30 milligrams (mg) (1 tablet of fezolinetant and 1 placebo tablet) once a day, fezolinetant 45 mg (2 tablets of fezolinetant) once a day or placebo (2 tablets) once a day. (Placebo was a dummy treatment that looked like medicine but did not have any medicine in it.) Women in this study were picked for 1 of the 3 study treatments by chance alone. The study participants took study treatment for 52 weeks.

This study was "double-blinded." That means that the study participants and the study doctors did not know who took which of the study treatments (fezolinetant 30 mg, fezolinetant 45 mg or placebo).

At weeks 2 and 4 and then once a month, the study participants went to the hospital or clinic for a check-up. They were asked about medications, side effects and how they felt. Other checks included physical exam and vital signs (heart rate, temperature and blood pressure). Blood and urine were collected for laboratory tests. At some study visits, study participants completed questionnaires that were about their quality of life. At the first and last study visits, they had a dual-energy x-ray absorptiometry (DXA for short) test done. To measure bone loss in the hips and spine, DXA created pictures of the inside of these areas with low-dose x-rays. (The dose was approximately one-tenth of the amount of a normal chest x-ray.) Study participants who still had their uterus had 2 more tests done at the first and last study visits. One of the 2 tests was endometrial biopsy. This test involved removing a small amount of tissue from the inside lining of the uterus. The tissue was then checked under a microscope. The other test was transvaginal ultrasound. It used sound waves to create pictures of the organs in the pelvis. The sound waves were transmitted by a probe (transducer), which was placed inside the vagina. Study participants might have had a screening mammogram done at the first and/or last study visit. A mammogram is an x-ray picture of the breasts used to screen for breast cancer. Study participants who did not had this test done in the last 12 months had it done at the first study visit. They had done at the last study visit if they were due for their screening mammogram and their own doctor agreed.

The last check-up at the hospital or clinic was at 3 weeks after the last dose of study treatment.

DETAILED DESCRIPTION:
This study consisted of a screening period and a 52 week treatment period. Safety follow up occurred 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥ 18 kg/m^2 and ≤ 38 kg/m^2.
* Subject must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

  * Spontaneous amenorrhea for ≥ 12 consecutive months
  * Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle stimulating hormone > 40 IU/L), or
  * Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit.
* Subject is seeking treatment for relief for VMS associated with menopause.
* Subject is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters; pulse rate and/or blood pressure; and ECG within the reference range for the population studied, or showing no clinically relevant deviations.
* Subject has documentation of a normal/negative or no clinically significant mammogram findings (obtained at screening or within the prior 12 months of study enrollment). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings.
* Subject is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and at week 52 end of treatment (EOT). For subjects who are withdrawn from the study prior to completion, a TVU should be collected at the early discontinuation (ED) visit.
* Subject is willing to undergo an endometrial biopsy at screening and at week 52 (EOT) or the ED visit for subjects who are withdrawn from the study prior to completion, and any time during the study in the case of uterine bleeding. The endometrial biopsy obtained at screening must be considered evaluable.
* Subject has documentation of a normal or not clinically significant Papanicolaou (Pap) test (or equivalent cervical cytology) within the previous 12 months or at screening.
* Subject has a negative urine pregnancy test at screening.
* Subject has a negative serology panel (i.e., negative hepatitis B surface antigen, negative hepatitis C virus antibody and negative human immunodeficiency virus antibody screens) at screening.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject uses a prohibited therapy (strong or moderate cytochrome P450 [CYP] 1A2 inhibitors, hormone replacement therapy [HRT], hormonal contraceptive, any treatment for VMS [prescription, over the counter or herbal]) or is not willing to wash out and discontinue such drugs for the full extent of the study.
* Subject has a known substance abuse or alcohol addiction within 6 months of screening.
* Subject has previous or current history of a malignant tumor, except for basal cell carcinoma.
* Subject's systolic blood pressure is ≥ 130 mmHg or diastolic blood pressure is ≥ 80 mmHg based on the average of 2 to 3 readings, on at least 2 different occasions within the screening period.

  * Subjects who do not meet these criteria may be re-assessed after initiation or review of antihypertensive measures.
  * Subjects with a medical history of hypertension can be enrolled once they are medically clear (stable and compliant).
* Subject has a history of severe allergy, hypersensitivity or intolerance to drugs in general, including the study drug and any of its excipients.
* Subject has an unacceptable result from the TVU assessment at screening, i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant finding.
* Subject has an endometrial biopsy confirming presence of disordered proliferative endometrium, endometrial hyperplasia, endometrial cancer, or other clinically significant findings at screening.
* Subject has a history within the last 6 months of undiagnosed uterine bleeding.
* Subject has a history of seizures or other convulsive disorders.
* Subject has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Subject has active liver disease, jaundice or elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP). Patients with mildly elevated ALT or AST up to 1.5 times the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Patients with mildly elevated ALP (up to 1.5 x ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Patients with Gilbert's syndrome with elevated total bilirubin may be enrolled as long as direct bilirubin, hemoglobin and reticulocytes are normal.
* Subject has creatinine > 1.5 x ULN; or estimated glomerular filtration rate using the Modification of Diet in Renal Disease formula ≤ 59 mL/min per 1.73 m^2 at the screening visit.
* Subject has a history of suicide attempt or suicidal behavior within the last 12 months or has suicidal ideation within the last 12 months (a response of "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide, as assessed at screening and at the time of visit 2 (randomization).
* Subject has previously been enrolled in a clinical trial with fezolinetant.
* Subject is participating concurrently in another interventional study or participated in an interventional study within 28 days prior to screening, or received any investigational drug within 28 days or within 5 half-lives prior to screening, whichever is longer.
* Subject is unable or unwilling to complete the study procedures.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has had a partial or full hysterectomy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1831 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (181):
- United States (141):
  - SEC Clinical Research, Andalusia, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Ensley, Alabama
  - Mesa Obstetricians and Gynecologists, Mesa, Arizona
  - Medpharmics LLC, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Visions Clinical Research - Tuscon, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Hope Research Institute, Canoga Park, California
  - Alliance Research Inc, Canoga Park, California
  - Marvel Clinical Research, Huntington Beach, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - National Research Institute - Panorama, Los Angeles, California
  - Excell Research, Oceanside, California
  - Clinical Trials Research, Sacramento, California
  - Northern California Research, Sacramento, California
  - Wake Research Associates, LLC, San Diego, California
  - Women's Healthcare Affiliates, San Diego, California
  - CITrials, Inc, Santa Ana, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Women's Medical Group of Upland, Upland, California
  - Bayview Research Group, Valley Village, California
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clincial Research Center LLC, Denver, Colorado
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Emerson Clinical Research institute, Washington D.C., District of Columbia
  - Olympian Clinical Research, Clearwater, Florida
  - Precision Clinical Research, Coral Springs, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Florida Medical Research, Gainesville, Florida
  - Vital Pharma Research Inc., Hialeah, Florida
  - Health Awareness, Jupiter, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Altus Research, Lake Worth, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Medical Research Center of Miami II, Miami, Florida
  - Medical Research Centers of South Florida, Inc., Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Spotlight research center, Miami, Florida
  - Med Research Of Florida, LLC, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Healthcare Clinical Data Inc, North Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Bioclinica Research, Orlando, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - Cornerstone Research Institute, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Sunset Point Medical Associates, Palm Harbor, Florida
  - Radiant Research, Pinellas Park, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Health Awareness, Port Saint Lucie, Florida
  - Precision Clinical Research, Sunrise, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Premier Medical Associates, The Villages, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - NuDirections Clinical Research, Duluth, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - WR-Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Georgia Clinical Research, Snellville, Georgia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - The Healing Sanctuary, LLC, Idaho Falls, Idaho
  - Womens Health USA, Inc., Champaign, Illinois
  - Affinity Clinical Research Institute, Oak Brook, Illinois
  - Investigators Research Group, Llc, Brownsburg, Indiana
  - MediSphere Medical Research, Evansville, Indiana
  - Cypress Medical Research Center, Wichita, Kansas
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Medpharmics, LLC, Metairie, Louisiana
  - Pharmasite Research Inc, Baltimore, Maryland
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Saginaw Valley Medical Research Group, Llc, Saginaw, Michigan
  - Montana Medical Research Inc, Missoula, Montana
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Clinical Research Center of Nevada (CRCN), Las Vegas, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Office Of Edmond Pack, Md, Las Vegas, Nevada
  - Dr.R. Garn Mabey, MD,Office Of, Las Vegas, Nevada
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Lawrence OBGYN Associates, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - Rochester Clinical Research, Inc., Rochester, New York
  - Circuit Clinical, West Seneca, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Carolina women's research and wellness center, Durham, North Carolina
  - Carolina Insitute for Clinical Research, Fayetteville, North Carolina
  - Unified Women's Clinical Research, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Unified Women's Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - CTI, Cincinnati, Ohio
  - Greater Cincinnati OB/GYN, Cincinnati, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Complete Healthcare For Women, Columbus, Ohio
  - Hwc Women's Research Center, Englewood, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - OB-GYN Associates, Erie, Pennsylvania
  - The Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Chattanooga GYN-Oncology, Chattanooga, Tennessee
  - WR Clinsearch, LLC, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - International Clinical Research, Murfreesboro, Tennessee
  - Tekton Research - Georgetown, Austin, Texas
  - Gadolin Research, LLC, Beaumont, Texas
  - DiscoveResarch, Inc., Bryan, Texas
  - Advances in Health, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - FMC Science, Lampasas, Texas
  - ClinRx Research, Plano, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Northeast Clinical Research Centers, Inc., Schertz, Texas
  - Excel Clinical Research, LLC, Sugar Land, Texas
  - EPIC Medical Research, Murray, Utah
  - Advanced Clinical Research-Old Farm OB/GYN (Utah), Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads Inc, Newport News, Virginia
  - Tidewater Clinical Research, Inc., Virginia Beach, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
- Canada (10):
  - Site CA15005, Brampton, Ontario
  - Site CA15006, Burlington, Ontario
  - Site CA15010, Sarnia, Ontario
  - Site CA15007, Toronto, Ontario
  - Site CA15012, Lévis, Quebec
  - Site CA15004, Point Claire, Quebec
  - Site CA15002, Québec, Quebec
  - Site CA15009, Québec, Quebec
  - Site CA15003, Sherbrooke, Quebec
  - Site CA15001, Victoriaville, Quebec
- Czechia (6):
  - Site CZ42008, Vodňany, Jihočeský kraj
  - Site CZ42001, Olomouc
  - Site CZ42003, Olomouc
  - Site CZ42010, Písek
  - Site CZ42009, Prague
  - Site CZ42005, Tábor
- Latvia (2):
  - Site LV37102, Riga
  - Site LV37101, Riga
- Poland (11):
  - Site PL48004, Bialystok
  - Site PL48005, Bydgoszcz
  - Site PL48002, Katowice
  - Site PL48019, Katowice
  - Site PL48006, Lublin
  - Site PL48014, Lublin
  - Site PL48016, Poznan
  - Site PL48010, Szczecin
  - Site PL48020, Warsaw
  - Site PL48003, Warsaw
  - Site PL48007, Warsaw
- Spain (2):
  - Site ES34005, Centelles
  - Site ES34002, Madrid
- Ukraine (2):
  - Site UA38004, Zaporizhzhya, Zaporizhzhia Oblast
  - Site UA38006, Kiev
- United Kingdom (7):
  - Site GB44003, Wokingham, Berkshire
  - Site GB44008, Sidcup, Kent
  - Site GB44005, Corby, Northamptonshire
  - Site GB44004, Kenilworth, Warwickshire
  - Site GB44006, Middlesex
  - Site GB44007, Romford
  - Site GB44001, Shipley

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kagan R, Cano A, Nappi RE, English ML, Mancuso S, Wu X, Ottery FD. Safety of Fezolinetant for Treatment of Moderate to Severe Vasomotor Symptoms Due to Menopause: Pooled Analysis of Three Randomized Phase 3 Studies. Adv Ther. 2025 Feb;42(2):1147-1164. doi: 10.1007/s12325-024-03073-8. Epub 2024 Dec 30. PMID 39739195
- [Derived] Neal-Perry G, Cano A, Lederman S, Nappi RE, Santoro N, Wolfman W, English M, Franklin C, Valluri U, Ottery FD. Safety of Fezolinetant for Vasomotor Symptoms Associated With Menopause: A Randomized Controlled Trial. Obstet Gynecol. 2023 Apr 1;141(4):737-747. doi: 10.1097/AOG.0000000000005114. Epub 2023 Mar 9. PMID 36897180
- See also: Link Description: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14543&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female participants aged ≥ 40 and ≤ 65 years seeking treatment for vasomotor symptoms (VMS) associated with menopause and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: Prior to randomization, participants had a screening period during which participants had transvaginal ultrasound, endometrial biopsy, dual-energy X-ray absorptiometry scan.
Groups:
- Placebo: Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, once daily (QD) for a of period of 52 Weeks.
- Fezolinetant 30 mg: Participants received fezolinetant 30 milligrams (mg) (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD for a period of 52 Weeks.
Period: Overall Study
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Started | 611 | 611 | 609
Treated | 610 | 611 | 609
Completed | 410 | 451 | 444
Not Completed | 201 | 160 | 165
Not completed — Adverse Event | 27 | 34 | 28
Not completed — Lost to Follow-up | 39 | 30 | 33
Not completed — Protocol Violation | 1 | 6 | 5
Not completed — Withdrawal by Subject | 119 | 79 | 85
Not completed — Miscellaneous | 14 | 11 | 14
Not completed — Participant did not receive study drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Fezolinetant 30 mg: Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD for a period of 52 Weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg | Total
Number analyzed (Participants) | 611 | 611 | 609 | 1831
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (4.8) | 54.7 (4.7) | 54.7 (4.8) | 54.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 611 | 611 | 609 | 1831
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 133 | 118 | 116 | 367
  Not Hispanic or Latino | 478 | 493 | 491 | 1462
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 2 | 8
  Asian | 8 | 8 | 13 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 92 | 114 | 110 | 316
  White | 502 | 479 | 479 | 1460
  More than one race | 6 | 6 | 4 | 16
  Unknown or Not Reported | 0 | 1 | 1 | 2
Smoking status [Number; unit: participants] — Participants with smoking status as current or former/never were reported.
  participants
    Current | 117 | 116 | 116 | 349
    Former/Never | 494 | 495 | 493 | 1482

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant administered a study drug, & which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign, symptom, or disease temporally associated with the use of medicinal product (MP) whether or not considered related to MP. An AE is considered "serious" if it results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inpatient hospitalization or leads to prolongation of hospitalization, hospitalization for treatment/observation/examination caused by AE is to be considered as serious, discontinuation due to increases in liver enzymes, other medically important events. A TEAE is defined as an AE observed after starting administration of study drug & 21 days after the last dose of study drug.
Time Frame: From first dose of study drug until 21 days after last dose of study drug (Up to 55 weeks)
Population: Safety analysis set (SAF) consisted of all randomized participants who took at least 1 dose of study intervention.
Measure: Number; unit: participants
Groups:
- Placebo: Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, QD for a period of 52 Weeks.
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 610 | 611 | 609
participants
  TEAE | 391 | 415 | 389
  Drug-Related TEAE | 106 | 94 | 110
  Serious TEAE | 14 | 20 | 23
  Drug-Related Serious TEAE | 1 | 0 | 0
  TEAE Leading to Death | 0 | 1 | 0
  Drug-Related TEAE Leading to Death | 0 | 0 | 0
  TEAE Leading to Withdrawal of Treatment | 26 | 34 | 28
  Drug-Related TEAE Leading to Withdrawal of Treatment | 16 | 16 | 17
  Death | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Mild, Moderate and Severe TEAE
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. A TEAE is defined as an AE observed after starting administration of the study drug and 21 days after the last dose of study drug. Severity of AE we were classified as Mild: No disruption of normal daily activities; Moderate: Affect normal daily activities; and Severe: Inability to perform daily activities.
Time Frame: From first dose of study drug until 21 days after last dose of study drug (Up to 55 weeks)
Population: SAF population
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 610 | 611 | 609
participants
  Mild | 180 | 215 | 195
  Moderate | 191 | 185 | 171
  Severe | 20 | 15 | 23

3. Primary Outcome: Percentage of Participants With Endometrial Hyperplasia
Description: Endometrial hyperplasia was confirmed from the endometrial biopsy report.
Time Frame: Baseline Up to 52 weeks
Population: Endometrial health set (EHS):All randomized participants who received at least 1 dose of study drug, had postbaseline (PB) biopsy done within 30 days after last dose, & had an acceptable biopsy at baseline (at least 1 endometrial biopsy (EB) with satisfactory tissue & no read of hyperplasia, disordered proliferative pattern or malignant) & had a satisfactory EB result after or on day 326 or had a PB final diagnosis of hyperplasia, disordered proliferative pattern or malignant prior to day 326.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 186 | 210 | 203
percentage of participants | 0 | 0 | 0.5

4. Primary Outcome: Percentage of Participants With Endometrial Cancer
Description: Endometrial cancer was confirmed from the endometrial biopsy report.
Time Frame: Baseline Up to 52 weeks
Population: Endometrial Health Set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 186 | 210 | 203
percentage of participants | 0 | 0.5 | 0

5. Secondary Outcome: Change From Baseline in Endometrial Thickness at Week 52
Description: Endometrial thicness was obtained from the transvaginal ultrasound. The endometrium was measured in the long axis or sagittal plane. The measurement was of the thickest echogenic area from 1 basal endometrial interface across the endometrial canal to the other basal surface.
Time Frame: Baseline and week 52
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 316 | 334 | 346
millimeter (mm) | -0.17 (2.35) | -0.15 (1.97) | -0.28 (2.30)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 30 mg; LSMeans (LSM), standard errors (SE), confidence intervals (CI); Test type: Superiority; p = 0.0604, ANCOVA — LSM, SE, CI, & p-values come from an analysis of covariance (ANCOVA) model with change from baseline at Week 52 timepoint as response, treatment & smoking status (current vs former/never) as fixed effects with baseline weight & baseline as covariate; LSMean difference = -0.08, 95% CI 2-sided [-0.36 to 0.21], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 45 mg; Test type: Superiority; p = 0.239, ANCOVA — The LSM, SE, CI, and p-values come from an ANCOVA model with change from baseline at the Week 52 timepoint as response, treatment and smoking status (current vs former/never) as fixed effects with baseline weight and baseline as covariates; LSMean difference = -0.17, 95% CI 2-sided [-0.45 to 0.11], Standard Error of Mean 0.14

6. Secondary Outcome: Percentage of Participants With Disordered Proliferative Endometrium
Description: Disordered proliferative endometrium was confirmed from the endometrial biopsy report.
Time Frame: Baseline Up to 52 weeks
Population: Endometrial Health Set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 186 | 210 | 203
percentage of participants | 2.2 | 1.4 | 0

7. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Hip at Week 52
Description: Changes in BMD hip was assessed by dual-energy X-ray absorptiometry (DXA) scan.
Time Frame: Baseline and week 52
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: gram per square centimeter (g/cm^2)
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 246 | 221 | 234
gram per square centimeter (g/cm^2)
  Hip (Femoral Neck) | -0.010 (0.033) | -0.001 (0.044) | -0.009 (0.033)
  Hip (Femur) | -0.011 (0.022) | -0.003 (0.041) | -0.008 (0.024)
  Hip (Trochanter) | -0.008 (0.027) | -0.001 (0.042) | -0.004 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Femoral Neck); Test type: Superiority; p = 0.029, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.007, 95% CI 2-sided [0.001 to 0.014], Standard Error of Mean 0.003
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Femoral Neck); Test type: Superiority; p = 0.867, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.001, 95% CI 2-sided [-0.006 to 0.007], Standard Error of Mean 0.003
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Femur); Test type: Superiority; p = 0.027, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.006, 95% CI 2-sided [0.001 to 0.012], Standard Error of Mean 0.003
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Femur); Test type: Superiority; p = 0.410, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.002, 95% CI 2-sided [-0.003 to 0.008], Standard Error of Mean 0.003
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Trochanter); Test type: Superiority; p = 0.087, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.005, 95% CI [-0.001 to 0.011], Standard Error of Mean 0.003
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Trochanter); Test type: Superiority; p = 0.259, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.003, 95% CI [-0.002 to 0.009], Standard Error of Mean 0.003

8. Secondary Outcome: Change From Baseline in Trabecular Bone Score (TBS) at Hip at Week 52
Description: TBS was a bone texture assessment that serves as a substitute for bone microarchitecture and predicts fracture risk independent of BMD and clinical risk factors. The DXA imaging was processed and analyzed as it would normally be and then evaluated using an automated algorithm to determine the TBS. T-score ≥1.350 was considered to be normal; T-score between 1.200 and 1.350 is considered to be consistent with partially degraded microarchitecture; and T-score ≤1.200 defines degraded microarchitecture.
Time Frame: Baseline and week 52
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: T-Score (Index)
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 246 | 221 | 234
T-Score (Index)
  Hip (Femoral Neck) | -0.078 (0.246) | -0.011 (0.372) | -0.073 (0.265)
  Hip (Femur) | -0.085 (0.192) | -0.024 (0.354) | -0.063 (0.192)
  Hip (Trochanter) | -0.071 (0.255) | -0.009 (0.426) | -0.036 (0.246)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Femoral Neck); Test type: Superiority; p = 0.079, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.048, 95% CI 2-sided [-0.006 to 0.102], Standard Error of Mean 0.027
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Femoral Neck); Test type: Superiority; p = 0.980, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.001, 95% CI 2-sided [-0.052 to 0.053], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Femur); Test type: Superiority; p = 0.042, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.048, 95% CI [0.002 to 0.094], Standard Error of Mean 0.023
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Femur); Test type: Superiority; p = 0.386, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.020, 95% CI [-0.025 to 0.065], Standard Error of Mean 0.023
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg; Hip (Trochanter); Test type: Superiority; p = 0.156, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.041, 95% CI [-0.016 to 0.099], Standard Error of Mean 0.029
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 45 mg; Hip (Trochanter); Test type: Superiority; p = 0.328, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.028, 95% CI 2-sided [-0.028 to 0.084], Standard Error of Mean 0.029

9. Secondary Outcome: Change From Baseline in BMD at Spine at Week 52
Description: Changes in BMD spine was assessed by DXA scan.
Time Frame: Baseline and week 52
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 253 | 225 | 242
g/cm^2 | -0.013 (0.035) | -0.010 (0.049) | -0.014 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 30 mg; Test type: Superiority; p = 0.497, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.002, 95% CI [-0.005 to 0.009], Standard Error of Mean 0.004
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 45 mg; Test type: Superiority; p = 0.878, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = -0.001, 95% CI [-0.007 to 0.006], Standard Error of Mean 0.004

10. Secondary Outcome: Change From Baseline in TBS at Spine at Week 52
Description: as for outcome 8
Time Frame: Baseline and week 52
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: T-Score (Index)
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 253 | 225 | 242
T-Score (Index) | -0.117 (0.296) | -0.084 (0.025) | -0.119 (0.298)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 30 mg; Test type: Superiority; p = 0.527, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = 0.020, 95% CI 2-sided [-0.042 to 0.082], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 45 mg; Test type: Superiority; p = 0.872, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LSMean difference = -0.005, 95% CI [-0.066 to 0.056], Standard Error of Mean 0.031

11. Secondary Outcome: Number of Participants With Suicidal Ideation and/or Behaviour as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS assessed the risk for suicidal behavior and suicide ideation. Participants responded as "Yes" or "No" 10 items. Suicidal ideation (1. Wish to be dead; 2. Non-specific active suicidal thoughts; 3. Active suicidal ideation with any methods (not plan) without intent to act; 4. Active suicidal ideation with some intent to act, without specific plan; 5. Active suicidal ideation with specific plan and intent; ). Suicidal behaviour (1. Preparatory acts or behavior 2. Aborted attempt 3. Interrupted attempt 4. Actual attempt 5. Completed suicide). Participants with 'Yes' to any one of the above 10 questions for suicidal ideation and behavior were reported.
Time Frame: Baseline, week 12, week 24, week 52 and follow-up (week 55)
Population: SAF population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 610 | 611 | 609
participants
  Baseline | 2 | 2 | 4
  Week 12: number analyzed (Participants) | 501 | 531 | 536
  Week 12 | 0 | 0 | 1
  Week 24: number analyzed (Participants) | 451 | 484 | 489
  Week 24 | 1 | 1 | 2
  Week 52: number analyzed (Participants) | 374 | 394 | 400
  Week 52 | 1 | 0 | 0
  Follow-up (Week 55): number analyzed (Participants) | 470 | 481 | 484
  Follow-up (Week 55) | 0 | 1 | 2

12. Secondary Outcome: Number of Participants With Self-injurious Behavior Without Suicidal Intent as Assessed by C-SSRS
Description: The C-SSRS assessed the risk for Self-injurious Behavior without Suicidal Intent. Question was asked "Has participant engaged in Non-Suicidal Self-Injurious Behavior?". Participants with 'yes' to the question were reported.
Time Frame: Baseline, week 12, week 24, week 52 and follow-up (week 55)
Population: SAF population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
Number analyzed (Participants) | 610 | 611 | 609
participants
  Baseline | 0 | 1 | 0
  Week 12: number analyzed (Participants) | 501 | 531 | 536
  Week 12 | 1 | 0 | 0
  Week 24: number analyzed (Participants) | 451 | 484 | 489
  Week 24 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 374 | 394 | 400
  Week 52 | 0 | 0 | 0
  Follow-up (Week 55): number analyzed (Participants) | 470 | 481 | 484
  Follow-up (Week 55) | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 21 days after last dose of study drug (Up to 55 weeks)
Description: SAF Population
Arm/Group | Placebo | Fezolinetant 30 mg | Fezolinetant 45 mg
All-Cause Mortality (participants affected / at risk) | 0/610 | 1/611 | 0/609
Serious Adverse Events (participants affected / at risk) | 14/610 | 20/611 | 23/609
Other Adverse Events (participants affected / at risk) | 90/610 | 86/611 | 78/609
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=610) | Fezolinetant 30 mg (N=611) | Fezolinetant 45 mg (N=609)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Alpha-1 antitrypsin deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=610) | Fezolinetant 30 mg (N=611) | Fezolinetant 45 mg (N=609)
COVID-19 (Infections and infestations) | 37 (37) | 38 (38) | 30 (30)
Headache (Nervous system disorders) | 56 (60) | 52 (57) | 54 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT04003389/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT04003389/SAP_001.pdf